CLINICAL TRIAL: NCT06175442
Title: Multicenter Non-randomized Controlled Retrospective Study of the Small Bowel Decompression Techniques Comparative Effectiveness in Patients With Benign Small Bowel Obstruction
Brief Title: Effectiveness of Small Bowel Decompression Techniques in Patients With Small Bowel Obstruction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: North-Western State Medical University named after I.I.Mechnikov (Other)
Responsible Party: Principal Investigator, Kotkov Pavel, Assistant of the Faculty Surgery Department in NWSMU, North-Western State Medical University named after I.I.Mechnikov
Other Study IDs: 17011993
Record Dates: First submitted 2023-12-06; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Small Bowel Obstruction; Small Bowel Obstruction Adhesion; Small-Bowel Obstruction Due to Volvulus; Hernia Incarcerated
Keywords: Acute intestinal obstruction, small bowel obstruction, nasointestinal tube, nasogastric tube

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Nasogastric tube only (I): Nasogastric intubation only will be the only method of intestinal decompression both intra- and postoperatively.
  Interventions: Device: Intraoperative intestinal decompression
- Short nasointestinal tube (IIA): Intraoperative intestinal decompression will be performed by placing the tube behind the ligament of Treitz and expressing the contents in the proximal direction or by total nasointestinal intubation with subsequent intraopertional tube withdrawal. Postoperative decompression will consist of the tube behind the ligament of Treitz.
  Interventions: Device: Intraoperative intestinal decompression
- Long nasointestinal tube intraoperative (IIB): Total intraoperative intubation of the small intestine followed by replacement with a nasogastric tube.
  Interventions: Device: Intraoperative intestinal decompression
- Long nasointestinal tube postoperative (IIC): Total intraoperative intubation of the small intestine with a long tube, which will persist in the postoperative period
  Interventions: Device: Intraoperative intestinal decompression

INTERVENTIONS:
Device: Intraoperative intestinal decompression — Insertion the tubes of various lengths (nasogastral, short and long nasointestinal) into the gastrointestinal tract during operations in patients with acute small intestinal obstruction

SUMMARY:
This study will compare results of different intestinal decompression techniques in patients with small bowel obstruction.

DETAILED DESCRIPTION:
Taking into account the large number of different variations of intestinal decompression methods, a comparative analysis will be carried out based on one comparison group (I) and three main ones (IA-B). The comparison criterion will be a group of patients with nasogastric drainage as the only method of the gastrointestinal tract decompression during surgery and in the postoperative period. In the main groups more active methods of intestinal decompression will be performed, including drainage of the initial parts of the small intestine or total intubation, both single-stage intraoperative and its extended version

ELIGIBILITY:
Inclusion Criteria:

* acute adhesive intestinal obstruction, including strangulation forms;
* incarcerated ventral hernias, accompanied by impaired intestinal passage;
* acute adhesive intestinal obstruction in the hernial sac;
* obstruction of the small intestine lumen with gallstones and other foreign bodies.

Exclusion Criteria:

* with peritonitis and other complicated surgical infection;
* operations with intestinal resection;
* patients after laparostomy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with benign forms of acute small intestinal obstruction and indications for the small intestine intubation: dilation of the the small intestine lumen above the level of a mechanical obstacle to 3.0 cm in diameter or more or the presence of intestinal paresis with the development of edema and microcirculatory disorders in intestinal wall.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
30-day postoperative mortality | 30 days after operation
  Number of patients, died during 30 days after the operation

SECONDARY OUTCOMES:
Postoperative complications | 30 days after operation
  Postoperative complications, defined according Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Locations (8):
- Russia (8):
  - Chelyabinsk regional clinical hospital, Chelyabinsk
  - City Clinical Hospital №4, Perm
  - North-Western State Medical University named after I. I. Mechnikov, Saint Petersburg
  - Saint-Petersburg I.I. Dzhanelidze Research Institute of Emergency Medicine, Saint Petersburg
  - St Petersburg State Budgetary Institution Of Health Care City Mariinskaya Hospital, Saint Petersburg
  - The City Hospital of the Holy Martyr Elizabeth, Saint Petersburg
  - State Healthcare Facility "City Clinical Emergency Hospital No 25", Volgograd
  - City Clinical Hospital No. 40, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No